CLINICAL TRIAL: NCT02453542
Title: Global Haemostatic Methods to Measure the Treatment Effect Following Administration of Bypassing Agents to Patients With Haemophilia With Inhibitors
Brief Title: Global Haemostatic Methods Following Administration of Bypassing Agents to Patients With Haemophilia With Inhibitors
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Roza Chaireti, MD, PhD, Karolinska Institutet
Other Study IDs: 202100-2973
Record Dates: First submitted 2015-05-17; First posted 2015-05-25 (Estimated); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Hemophilia
Keywords: hemophilia; inhibitors; thrombin
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Background

The treatment of haemophilia A and B has been revolutionized by the use of factor concentrate, both as prophylaxis and to treat bleeding episodes (on-demand treatment). However, despite its advantages, repeated treatment with factor concentrate can lead to development of inhibitors (antibodies) towards the coagulation factor in the concentrate. Another patient group in which the bleeding symptoms are difficult to treat because of inhibitors towards coagulation factors, most commonly FVIII, is patients with acquired haemophilia. Patients with high antibody titers exhibit a deficient or no response to factor concentrates and usually need treatment with bypassing agents, namely factor eight inhibitor bypassing agent (FEIBA®, Baxter) och recombinant activated factor VII (rFVIIa, Novo-Seven®, Novo Nordisk). The effect of the treatment cannot be accurately monitored by traditional coagulation tests.

The aim of the study is to evaluate the utility of the global haemostatic methods in patients with haemophilia with inhibitors. The objective is to improve the monitoring of the treatment effect and thus increase the safety of the patient and the effectiveness of the treatment.

Patients and methods

Patients

The primary cohort will consist of fifteen patients with inherited haemophilia with inhibitors as well as five adult patients with acquired haemophilia who are followed up at the Coagulation Department of the Karolinska University Hospital, Stockholm, Sweden.

Blood samples will be collected from those patients at specific time points (see Design of the study) during the course of two years (for each patient). The treatment (type, dose, duration) will be determined by the treating physician.

Methods (selection)

* Thrombin generation (Calibrated Automated Thrombogram, CAT® and a commercial kit from Siemens®).
* Overall haemostatic potential (OHP)

Design of the study

Timeframe for blood sampling: i) baseline (inclusion in the study), and ii) prior and after administration of bypassing agents to either treat bleeding symptoms or before an invasive procedure or as prophylaxis.

Data analysis

The variations in coagulation markers measured as described above (Methods) will be associated to the clinical symptoms (bleeding), the level of coagulation factors (if measurable) and the titers of the inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* meets the study population description

Exclusion Criteria:

* no informed consent age<7 years

Min Age: 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Fifteen patients (adults and children) with hereditary haemophilia with inhibitors.
  Five patients (adults) with acquired haemophilia
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-03-01 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Changes in coagulation markers, such as thrombin generation markers (Endogenous Thrombin Potential in nano molar thrombin*minute and peak thrombin in nano molar and fibrin aggregation curves, following administration of bypassing agents.) composite | participants will be followed up for up to 2 years following inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Roza Chaireti, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Solna, Stockholm County, Sweden